CLINICAL TRIAL: NCT05250531
Title: Efficacy of Telerehabilitation and Multicomponent Therapy in Women With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Multicomponent Therapy With Telerehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, DIREN OZER OZBEY, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Istanbul University,Istanbul
Record Dates: First submitted 2022-01-24; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia
Keywords: telerehabilitation; multicomponent therapy; psychotherapy; pain; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Experimental): 33 patients in the multicomponent treatment group selected to group 1 (G1) will be treated with telerehabilitation for a total of 6 sessions of two hours once a week for 3 weeks. After 1 month, one more session will be applied for a two-hour follow-up and sustainability.
  Interventions: Behavioral: multicomponent therapy
- GROUP 2 (Active Comparator): As a control group, 33 patients selected to Group 2 (G2) will be given exercise and training with telerehabilitation.
  Interventions: Behavioral: multicomponent therapy

INTERVENTIONS:
Behavioral: multicomponent therapy — patient education,Exercise training,Private Psychotherapy,relaxation

SUMMARY:
In this prospective, randomized study, our aim was to evaluate the comprehensive multicomponent treatment of fibromyalgia women with telerehabilitation, including "patient education, special psychotherapy/psychosocial intervention, and exercise including relaxation exercises". Does it differ in terms of reduction and functionality?

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be randomized into two groups by computer program after being numbered according to the order of application. 33 patients in the multicomponent treatment group selected to group 1 (G1) will be treated with telerehabilitation for a total of 6 sessions of two hours once a week for 3 weeks. After 1 month, one more session will be applied for a two-hour follow-up and sustainability. As a control group, 33 patients selected to Group 2 (G2) will be given exercise and training with telerehabilitation.

Patients to whom a multicomponent treatment program will be applied will be included in the program in groups of 10. The presentations will be prepared as power-point presentations and will be presented to the patients online with telerehabilitation.

Interventions to be applied in the multicomponent treatment protocol:

1. Patient education
2. Exercise training
3. Private Psychotherapy
4. Relaxation

ELIGIBILITY:
Inclusion Criteria:

1. Women
2. Symptom persistence for more than 3 months
3. Pervasive Network Scale Score >7 and Symptom Severity Score >5 according to 2016 ACR criteria
4. Symptom Severity Score of >9 and Diffuse Pain Scale Score between 4-6 according to 2016 ACR criteria
5. Getting a high (11 and above) score on the Hospital Anxiety and Depression Scale
6. Having the opportunity to participate in the applications online
7. No change in the medical treatment he received for fibromyalgia syndrome during the study period
8. Those between the ages of 18-55

Exclusion Criteria:

1. Patients with endocrine, neuromuscular, infectious and inflammatory rheumatological diseases
2. Patients with liver or kidney disease
3. Patients with malignancy
4. Patients with a history of severe trauma
5. Patients with severe psychiatric illness
6. Patients with serious physical comorbidities
7. The illiterate
8. Known central nervous system or peripheral nervous system disease, progressive neurological deficit
9. Peripheral venous insufficiency, coagulopathies and anticoagulant drug use
10. Serious cardiovascular pathologies
11. Loss of sensation, loss of position sense, unhealed fracture or open surgical wound
12. Pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — effect of gender difference on intervention outcomes
Enrollment: 66 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
change in The Revised Fibromyalgia Impact Questionnaire (FIQR) | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  The fibromyalgia impact questionnaire was developed from information gathered from patient reports, functional status tools, and clinical observations. This questionnaire measures physical function, work status (days off and work difficulty), depression, anxiety, morning fatigue, pain, stiffness, fatigue, and well-being in the past week.

SECONDARY OUTCOMES:
change in Jenkins Sleep Evaluation Questionnaire (JSEQ) | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  It is important to evaluate and treat sleep problems. It consists of four items that evaluate sleep problems in the last four weeks. It is a simple, time-consuming and easily calculated sleep assessment tool that can be used in fibromyalgia patients.
change in The Fatigue Severity Scale (FSS) | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  It consists of nine items that measure the severity of the patients' fatigue symptoms in the last week. It assesses the prevalence and severity of fatigue, the management of affected patients, and the monitoring of disease-related fatigue.
change in Visual Analogue Scale (VAS) | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  Pain will be evaluated with the Visual Analogue Scale (VAS). The numerical value obtained by measuring in millimeters will show the patient's pain intensity (0 = no pain, 10 = most severe pain). The patient will be asked about the average of the pain intensity felt in the last week.
change in ICF Core Set for Chronic Widespread Pain | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  It was aimed to determine the functional characteristics of the patients, the impairments in body functions, activity limitations and participation limitations, and the facilitating or inhibiting effects of environmental factors.
change in The Central Sensitization (CSI) Inventory | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  It is a scale used to detect patients with symptoms related to central sensitization or types of central sensitization syndrome such as fibromyalgia, temporomandibular joint disease, tension-type headache, migraine.
change in hospital anxiety and depression scale | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  It is a self-report scale consisting of 14 items. Single items provide an assessment of anxiety and dual items of depression. It is used in the evaluation of patients with physical health since it does not contain physical symptoms.
change in Short Form-36 (SF-36) | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  Quality of life will be measured with Short Form-36 (Short Form-36, SF-36). SF-36 is one of the most widely used criteria among generic criteria. It is a valid and frequently used criterion for assessing quality of life. It is not specific to any age, disease or treatment group. It includes general health concepts. It was developed for use in clinical practice and research. It includes 36 questions on eight subscales: physical function, physical role difficulty, body pain, general health, vitality, social function, emotional role difficulty, and mental health.
change in Pain Coping Inventory (PCI) | Baseline (before intervention), 1 month after intervention, 3 months after the intervention
  It was developed by Kraaimaat and Evers (2003) in order to determine the behavioral and cognitive strategies used by chronic pain patients to cope with pain. It consists of six sub-dimensions and 22 items. The lowest score that can be obtained from all sub-dimensions of the questionnaire, which is evaluated with a 4-point Likert type, is one and the highest score is four. Sub-dimensions are scored by dividing by the number of items.
change in Pain Self Efficacy Questionnaire-2 (PSEQ-2) | Baseline (before intervention), after a month intervention, after 3 month the intervention
  It is stated that self-efficacy for coping with pain can also be measured with a two-item short form. The high score obtained from the questionnaire evaluated with a five-point Likert-type scale indicates that the individuals' self-efficacy regarding pain has increased. A minimum of one and a maximum of five points are taken from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Diren Ozer Ozbey, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No